CLINICAL TRIAL: NCT04893954
Title: Prospective Study on the Consequences of Weight Loss After Bariatric Surgery on Obese Patients' Spine : Effects on Low Back Pain, Sagittal Alignment and Lipomatosis.
Brief Title: Prospective Study on the Consequences of Weight Loss After Bariatric Surgery on Obese Patients' Spine.
Acronym: SPINOB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Sauver La Vie (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP201602
Record Dates: First submitted 2021-02-24; First posted 2021-05-20 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain in Obese Patients After Important Weight Loss
Keywords: Bariatric; Spine; Obese; Low back pain; Sagittal alignment; Lipomatosis
MeSH Terms: conditions — Obesity; Low Back Pain; Lipomatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Obese patients (Other)
  Interventions: Diagnostic Test: Full Spine Radiography; Diagnostic Test: Lumbar spine MRI

INTERVENTIONS:
Diagnostic Test: Full Spine Radiography — Full Spine Radiography
Diagnostic Test: Lumbar spine MRI — Lumbar spine MRI

SUMMARY:
The purpose of this study is to determine how an important weight loss after bariatric surgery affects obese patients ' spine, and the effects it has on low back pain, sagittal alignment and lipomatosis .

DETAILED DESCRIPTION:
Obesity and back pain are massive public health problems, and the relationship between the two has not been described and studied. However, the investigators have also observed that many ex-obese patients still suffer from back and leg pain after an important weight loss.

The aim of this study is to measure the effect of weight loss on back pain, and to find out what parameters can explain such modifications (increasing or decreasing back pain).

The investigators will study clinical parameters, as well as radiological (to measure the effect of weight loss on spine sagittal alignment) and MRI (to measure lipomatosis, which is a fat epidural accumulation, responsible for nerve compression and therefore back and leg pain).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* BMI > 40 or BMI > 35 with comorbidities due to obesity ( criteria for bariatric surgery)
* Follow up in Pompidou's Hospital Nutrition service
* Bariatric surgery intervention ( Sleeve gastrectomy or By pass)
* Follow up possible for one year or more
* Being covered by French social insurance
* Consent to participate in the study

Exclusion Criteria:

* History of spine surgery
* Bariatric surgery postoperative complication
* Non mastering of french language
* MRI contraindication
* Patient under legal protection ( e.g. guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Oswestry disability Index (ODI) | 1 year postoperative
  Clinical score to evaluate low back pain vs Preoperative evaluation
Oswestry disability Index (ODI) | 2 years postoperative
  Clinical score to evaluate low back pain vs Preoperative evaluation

SECONDARY OUTCOMES:
Oswestry disability Index (ODI) | 6 months postoperative
  Clinical score to evaluate low back pain vs Preoperative evaluation
Sagittal alignment | 6 months postoperative
  Radiologic measurement of spine parameters vs Preoperative evaluation
Sagittal alignment | 1 year postoperative
  Radiologic measurement of spine parameters vs Preoperative evaluation
Sagittal alignment | 2 years postoperative
  Radiologic measurement of spine parameters vs Preoperative evaluation
Disc degeneration | 6 months postoperative
  MRI evaluation vs Preoperative evaluation
Disc degeneration | 1 year postoperative
  MRI evaluation vs Preoperative evaluation
Disc degeneration | 2 years postoperative
  MRI evaluation vs Preoperative evaluation
Lipomatosis | 6 months postoperative
  MRI evaluation of lumbar epidural fat accumulation vs Preoperative evaluation
Lipomatosis | 1 year postoperative
  MRI evaluation of lumbar epidural fat accumulation vs Preoperative evaluation
Lipomatosis | 2 years postoperative
  MRI evaluation of lumbar epidural fat accumulation vs Preoperative evaluation
Visual Analog Scale (VAS) | 6 months postoperative
  Clinical score to evaluate low back pain vs Preoperative evaluation
Visual Analog Scale (VAS) | 1 year postoperative
  Clinical score to evaluate low back pain vs Preoperative evaluation
Visual Analog Scale (VAS) | 2 years postoperative
  Clinical score to evaluate low back pain vs Preoperative evaluation
Neck disability Index (NDI) | 6 months postoperative
  clinical score to evaluate neck pain vs Preoperative evaluation
Neck disability Index (NDI) | 1 year postoperative
  clinical score to evaluate neck pain vs Preoperative evaluation
Neck disability Index (NDI) | 2 years postoperative
  clinical score to evaluate neck pain vs Preoperative evaluation
Short Form 12 (SF12) | 6 months postoperative
  Score to evaluate quality of life vs Preoperative evaluation
Short Form 12 (SF12) | 1 year postoperative
  Score to evaluate quality of life vs Preoperative evaluation
Short Form 12 (SF12) | 2 years postoperative
  Score to evaluate quality of life vs Preoperative evaluation
Hospital anxiety and depression (HAD) scale | 6 months postoperative
  Score to evaluate depression vs Preoperative evaluation
Hospital anxiety and depression (HAD) scale | 1 year postoperative
  Score to evaluate depression vs Preoperative evaluation
Hospital anxiety and depression (HAD) scale | 2 years postoperative
  Score to evaluate depression vs Preoperative evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle FERRERO, MD, PHD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Briggs MS, Givens DL, Schmitt LC, Taylor CA. Relations of C-reactive protein and obesity to the prevalence and the odds of reporting low back pain. Arch Phys Med Rehabil. 2013 Apr;94(4):745-52. doi: 10.1016/j.apmr.2012.11.026. Epub 2012 Nov 24. PMID 23187041
- [Background] Khoueir P, Black MH, Crookes PF, Kaufman HS, Katkhouda N, Wang MY. Prospective assessment of axial back pain symptoms before and after bariatric weight reduction surgery. Spine J. 2009 Jun;9(6):454-63. doi: 10.1016/j.spinee.2009.02.003. Epub 2009 Apr 8. PMID 19356988
- [Background] Koulischer S, Cadiere B, Cadiere GB, Fabeck L. [Evolution of low back pain after bariatric surgery]. Rev Med Brux. 2015 May-Jun;36(3):147-51. French. PMID 26372975
- [Background] de Mello AP, Martins GCDS, Heringer AR, Gamallo RB, Martins Filho LFDS, de Abreu AV, Carvalho ACP, Gama MP. Back pain and sagittal spine alignment in obese patients eligible for bariatric surgery. Eur Spine J. 2019 May;28(5):967-975. doi: 10.1007/s00586-019-05935-0. Epub 2019 Mar 15. PMID 30877387
- [Background] Beckworth WJ, McCarty EJ, Garcia-Corrada JE, Holbrook JF. Epidural Lipomatosis and Associated Spinal Stenosis-The Impact of Weight Loss: A Case Report. Am J Lifestyle Med. 2017 Jan 12;11(6):511-514. doi: 10.1177/1559827616686764. eCollection 2017 Nov-Dec. PMID 30202377
- [Background] Joaquim AF, Helvie P, Patel AA. Bariatric Surgery and Low Back Pain: A Systematic Literature Review. Global Spine J. 2020 Feb;10(1):102-110. doi: 10.1177/2192568219826935. Epub 2019 Feb 5. PMID 32002354